CLINICAL TRIAL: NCT02186925
Title: A Prospective Study of Clinical Factors Affecting Disease Progression and Treatment Results of Patients With Tumors of the Prostate, Bladder and Kidney.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ren001
Record Dates: First submitted 2014-07-02; First posted 2014-07-10 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2014-07

CONDITIONS: Kidney Cancer; Prostate Cancer; Bladder Cancer
Keywords: Kidney Cancer; Prostate Cancer; Bladder Cancer
MeSH Terms: conditions — Kidney Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bladder, Kidney and Prostate Cancer Patients

SUMMARY:
Identifying clinical factors such as medication, background diseases and blood tests that effect the course of disease in cancer patients can help physicians to better decide on the patient's treatment plan. The study seeks to identify and analyze relevant clinical factors that effect the course of the disease and the results of treatment in patients with cancers of the prostate, bladder and kidney.

ELIGIBILITY:
Inclusion Criteria:

* All patients with prostate, bladder or kidney cancer that are being treated at the Meir Medical Center and are over 18 years of age.

Exclusion Criteria:

* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from kidney, bladder or prostate cancer who are being treated at the Meir Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-08; Primary Completion 2019-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 5 years
  Univariate analysis will be used to assess the effects of clinical factors on progression free survival.

SECONDARY OUTCOMES:
Patient overall survival | 5 years
  Univariate analysis will be used to assess the effects of clinical factors on overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Daneil Kejzman, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kvar Saba, Israel